CLINICAL TRIAL: NCT00004669
Title: Phase II Pilot Study of Early Cortisol Replacement to Prevent Bronchopulmonary Dysplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Penn State University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Prevention
Other Study IDs: 199/12016; PENN-420633
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: bronchopulmonary dysplasia; cardiovascular and respiratory diseases; neonatal disorders; rare disease
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Respiratory Tract Diseases; Infant, Newborn, Diseases; Rare Diseases | interventions — Hydrocortisone

INTERVENTIONS:
Drug: hydrocortisone

SUMMARY:
OBJECTIVES: I. Estimate the efficacy of cortisol replacement therapy during the first 12 days of life for prevention of bronchopulmonary dysplasia.

II. Estimate the effect of cortisol replacement therapy on the signs of acute adrenal insufficiency.

III. Evaluate the effects of cortisol replacement therapy on adrenal hormone concentrations and on the ability of the adrenal gland to respond to ACTH.

IV. Determine the effect of this replacement therapy on markers of inflammation in lung lavage fluid and peripheral blood leukocytes.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled study. Hydrocortisone therapy IV or placebo begins no later than 48 hours after birth and continues every 12 hours for 12 days. Hydrocortisone is given at 2-4 times the basal cortisol secretion rate.

Tracheal lavage on intubated babies is performed at start of study and on day 4 of life to assess concentrations of inflammatory markers.

If larger babies show appropriate response to ACTH by 15-17 days and the less mature babies show a decreased response, then a longer course of therapy is proposed for future studies.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* At risk for development of bronchopulmonary dysplasia

--Patient Characteristics--

* Hematopoietic: No congenital sepsis
* Hepatic: No structural defect of liver
* Renal: No agenesis or structural defect of a kidney
* Cardiovascular: No structural defect of the heart
* Metabolic: No diabetic mothers (e.g., preexisting insulin dependent, noninsulin dependent, and gestational diabetes)
* Pulmonary: No structural defect of the lung
* Other: Newborn birth weight must be 500 to 999 g and have endotracheal tubes in place at 12 hours of age Eligible if treatment can be given before 48 hours of postnatal life No major congenital anomaly causing significant defect in major organ system

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40
Dates: Start 1996-06

CONTACTS AND LOCATIONS:
Overall Officials: Kristi L. Watterberg, Study Chair — Penn State University